CLINICAL TRIAL: NCT04785586
Title: Effective Weight Maintenance for the Working Age - the Effectivity and Adherence of Three Web-based Weight Maintenance Interventions
Brief Title: Effective Weight Maintenance for the Working Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Occupational Health Helsinki (Unknown); University of Helsinki (Other)
Responsible Party: Principal Investigator, Kirsi Pietiläinen, Professor in Clinical Metabolism, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200379
Record Dates: First submitted 2021-02-10; First posted 2021-03-08 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Obesity
Keywords: Weight management; Occupational health
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The patients are randomized into three groups all of which include the HealthyWeightCoaching (HWC) platform. In addition, group 1 will be offered three individual face-to-face sessions via video and group 2 three group face-to-face sessions via video. Group 3 acts as the control group offering the basic HWC protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual (Experimental): HWC protocol + three individual "face-to-face" sessions via video
  Interventions: Behavioral: Healthy Weight Coaching; Behavioral: Individual meetings
- Group (Experimental): HWC protocol + three "face-to-face" group sessions via video
  Interventions: Behavioral: Healthy Weight Coaching; Behavioral: Group meetings
- Control (Active Comparator): Standard HWC protocol
  Interventions: Behavioral: Healthy Weight Coaching

INTERVENTIONS:
Behavioral: Healthy Weight Coaching — Lifestyle intervention based on Healthy Weight Coaching (HWC) is a 52 week long web-based weight loss program consisting of weekly modules, exercises, peer support, and one-on-one coaching. It encompasses themes such as diet, physical activity, coping with stress, sleep, and general health.
Behavioral: Individual meetings — Individual sessions via video, offered to the participant at three (3) different time points during the 12 month intervention.
  Arms: Individual
Behavioral: Group meetings — Group sessions via video, offered to the participant at three (3) different time points during the 12 month intervention.
  Arms: Group

SUMMARY:
This study aims to compare the effectiveness and adherence of three web-based weight management interventions, all based on the HealthyWeightCoaching (HWC) within a HealthyWeightHub.fi (HWH) platform. HWC is a 12-month web-based intervention including information and exercises to promote weight loss. Each patient is allocated a personal coach to encourage progress on the platform.

In the current setting, the investigators study how minimal added support will affect the effectiveness and adherence of the web-based program. The patients are randomized into three groups all of which include the HWC platform. In addition, group 1 will be offered three individual face-to-face sessions via video and group 2 three group face-to-face sessions via video. Group 3 acts as the control group offering the basic HWC protocol.

The patients (target n=120) are enrolled from the occupational health of the city of Helsinki.

DETAILED DESCRIPTION:
Obesity is one of the major public health problems globally, affecting an ever-increasing proportion of working age adults. In addition of increasing the risk of many obesity-associated diseases, obesity is associated to impaired ability to work, making it a relevant occupational health concern. Treatment of obesity requires long-term interventions, but nevertheless, it is challenging to provide long-term treatment when resources in real-life health care systems are limited. To that need, new cost-effective and accessible intervention methods are created. One of these is the a real-life web-based obesity management program HealthyWeightCoaching (HWC).

HWC has shown promising results in obesity management, but alike in other fully virtual interventions, one of the challenges has been adherence. Creating hybrid-models by addition of face-to-face contacts to the web-based structure, has been shown to improve adherence and therefore the effectiveness of the intervention. However, data on hybrid interventions for weight management is still scarce and calls for further research.

In the current setting, the investigators study how minimal added support will affect the effectiveness and adherence of the web-based program. The patients are randomized into three groups all of which include the HWC platform. In addition, group 1 will be offered three individual face-to-face sessions via video and group 2 three group face-to-face sessions via video. Group 3 acts as the control group offering the basic HWC protocol.

Data on health and lifestyle are collected at 0, 6, 12 month time points. The 12-month intervention is followed by a 5 year monitoring period. The data collection includes questionnaires, measurements and laboratory tests.

The patients (target n=120) are enrolled from the occupational health of the city of Helsinki. The participation is free for the patient.

ELIGIBILITY:
Inclusion Criteria:

* working age
* body mass index (BMI) 30-40 kg/ m²
* the possibility to use a computer and /or a smartphone with access to the internet
* willingness to participate in the treatment program
* sufficient Finnish language

Exclusion Criteria:

* diagnosed severe illness (incl. mental illnesses)
* pregnancy or breastfeeding
* simultaneous participation in another weight loss program
* remarkable changes in weight (+/- 5kg) in the past 3 months
* bariatric operation (past or upcoming)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent of weight loss | baseline to 24 months
  Mean weight change in percent

SECONDARY OUTCOMES:
Categorical weight loss | baseline to 24 months
  Percent of patients achieving 3-4.9 percent, 5-9.9 percent and >10 percent weight loss
Psychological Flexibility | baseline to 24 months
  Psychological flexibility is assessed by the Acceptance and Action Questionnaire for Weight (AAQW). It is a 22-item, Likert-type scale that measures acceptance of weight related thoughts and feelings with valued actions. Theoretical range of the overall score is 22-154, higher scores indicating worse outcome.
Eating behaviour | baseline to 24 months
  Eating behavior is assessed by the Three Factor Eating Questionnaire (TFEQ). The Three-Factor Eating Questionnaire (TFEQ), a valid 51-item measure of restraint, disinhibition, and hunger subscales. Theoretical range of the overall score is 0-51, higher scores indicating worse outcome.
Perceived working ability | baseline to 24 months
  Perceived working ability is assessed by a simple "How able do you feel like to manage your job at the moment". The score is measured by a ten point scale (1-10), higher score indicating better outcome.
Glucose metabolism | baseline to 24 months
  Concentration of fasting glucose and HbaA1c in a blood sample
Lipid metabolism | baseline to 24 months
  Concentration of fasting cholesterol (HDL, LDL, trigly) in a blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Siniriikka Männistö, Psy.M./MHS, Study Director — Occupational Health Helsinki
Locations (1):
- Occupational Health Helsinki, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mannisto SA, Pietilainen KH, Muotka J, Suojanen LU, Lappalainen R, Korpela R. Coach-Assisted eHealth With Group or Individual Support for Employees With Obesity: Randomized Controlled Trial on Weight, Body Composition, and Health Metrics. J Med Internet Res. 2025 Mar 12;27:e60436. doi: 10.2196/60436. PMID 40073400